CLINICAL TRIAL: NCT01806623
Title: A Multicenter Open-label Non-comparative Study Of Fluconazole For The Treatment Of Vulvovaginal Candidiasis.
Brief Title: The Study Of Fluconazole For Vulvovaginal Candidiasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A0561023
Record Dates: First submitted 2013-01-28; First posted 2013-03-07 (Estimated); Results first posted 2014-12-03 (Estimated); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Vulvovaginal Candidiasis
MeSH Terms: conditions — Candidiasis, Vulvovaginal | interventions — Fluconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fluconazole (Experimental)
  Interventions: Drug: Fluconazole

INTERVENTIONS:
Drug: Fluconazole — Single oral dose of 150mg Fluconazole

SUMMARY:
As for the indication of vulvovaginal candidiasis, a single oral administration of fluconazole 150 mg has been approved and is recommended by guidelines overseas. However in Japan oral therapy with antifungal triazole such as Fluconazole has not been approved, and topical therapies such as vaginal tablets, pessary and cream are used clinically. The purpose of this trial is to confirm the efficacy and safety of single oral administration of fluconazole 150 mg for the treatment of vulvovaginal candidiasis in Japanese patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical symptoms and signs of vulvovaginal candidiasis.
* Patients tested positive for Candida by fungal culture.
* Patients who can agree not to have intercourse up to 28 days after dosing.

Exclusion Criteria:

* Patients with a history of hypersensitivity to fluconazole.
* Patients with severe renal dysfunction.
* Patients with liver disorder.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2013-03-05 (Actual); Primary Completion 2013-11-22 (Actual); Study Completion 2013-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (10):
- Japan (10):
  - Ai WOMEN'S CLINIC, Asahikawa, Hokkaido
  - Shirokane Ladies' Clinic, Minato-ku, Tokyo
  - Takane Medical Clinic, Shinagawa-ku, Tokyo
  - Suzuran Clinic, Suginami-ku, Tokyo
  - Mori Ladies Clinic, Fukuoka
  - IZUMI Ladies' Clinic, Gifu
  - Tetsu-Nakamura Obstetrics and Gynecology Department Internal Medicine, Kagoshima
  - Women's Clinic Kamimura, Okayama
  - Sutou Ladies Clinic, Osaka
  - Hayakawa Clinic, Osaka

REFERENCES:
- [Derived] Mikamo H, Matsumizu M, Nakazuru Y, Okayama A, Nagashima M. Efficacy and safety of a single oral 150 mg dose of fluconazole for the treatment of vulvovaginal candidiasis in Japan. J Infect Chemother. 2015 Jul;21(7):520-6. doi: 10.1016/j.jiac.2015.03.011. Epub 2015 Mar 30. PMID 25887336
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0561023&StudyName=The%20Study%20Of%20Fluconazole%20For%20Vulvovaginal%20Candidiasis

RESULTS

PARTICIPANT FLOW:
Groups:
- Fluconazole: Three fluconazole 50 mg capsules were orally administered once on the first day of the treatment
Period: Overall Study
Arm/Group | Fluconazole
Started | 157
Completed | 99
Not Completed | 58
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1
Not completed — Did not meet the inclusion criteria | 56

BASELINE CHARACTERISTICS:
Arm/Group | Fluconazole
Number analyzed (Participants) | 157
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.8 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 157
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Therapeutic Outcome: Response Rate
Description: Therapeutic outcome was determined by combination of clinical efficacy and mycological efficacy for each participant as Effective, Ineffective or Indeterminate. The therapeutic outcome was considered as Effective when the clinical efficacy was Cure and the mycological efficacy was Eradication.
  Primary evaluation of therapeutic outcome was on Day 28.
  Response rate was calculated based on the following formula, "the number of participants assessed as effective" over "total participants excluding ones assessed as indeterminate" multiplied by 100.
Time Frame: Day 7, Day 14 and Day 28
Population: The modified-Intent to Treat (m-ITT) included participants with vulvovaginal candidiasis who received the investigational products, who tested positive for Candida in the vulva and/or vagina at Day 1 (before dosing), and whose clinical efficacy was evaluated.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fluconazole
Number analyzed (Participants) | 102
percentage of participants
  Day 7 (n=95) | 33.7 [24.2 to 44.3]
  Day 14 (n=100) | 54.2 [43.7 to 64.4]
  Day 28 (n=102) | 74.7 [65.0 to 82.9]

2. Secondary Outcome: Clinical Efficacy: Cure Rate
Description: Scores of severity in signs and symptoms at each observation dates were compared with those before the treatment and the clinical efficacy was determined as Cure (the clinical symptom disappeared), Improvement (the clinical symptom was improved: the total score of clinical symptom was reduced relative to the total score before the treatment), Failure (the criteria for Cure and Improvement were not met, or other systemic antifungal drugs or local antifungal drugs were administered for the treatment of the disease to be examined) or Indeterminate (efficacy for each item was not determined for the reasons including failure to conduct the test, or other systemic antifungal agents or local antifungal drugs were administered for the treatment of infections other than the disease to be examined).
  Cure rate was calculated based on the following formula, "the number of participants assessed as Cure" over "total participants excluding ones assessed as Indeterminate" multiplied by 100.
Time Frame: Day 7, Day 14 and Day 28
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fluconazole
Number analyzed (Participants) | 102
percentage of participants
  Day 7 (n=99) | 34.8 [25.1 to 45.4]
  Day 14 (n=101) | 57.3 [46.8 to 67.3]
  Day 28 (n=102) | 81.6 [72.5 to 88.7]

3. Secondary Outcome: Clinical Efficacy: Cure and Improvement Rate
Description: Scores of severity in signs and symptoms on each observation dates are compared with those before the treatment and the clinical efficacy is determined as Cure (the clinical symptom disappeared), Improvement (the clinical symptom was improved), Failure (the criteria for Cure and Improvement were not met, or other systemic antifungal drugs or local antifungal drugs were administered for the treatment of the disease to be examined) or Indeterminate (efficacy for each item was not determined for the reasons including failure to conduct the test, or other systemic antifungal agents or local antifungal drugs were administered for the treatment of infections other than the disease to be examined).
  Cure and improvement rate was calculated based on the following formula, "the number of participants assessed as Cure or Improvement" over "total participants excluding ones assessed as Indeterminate" multiplied by 100.
Time Frame: Day 7, Day 14 and Day 28
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fluconazole
Number analyzed (Participants) | 102
percentage of participants
  Day 7 (n=99) | 100.0 [96.1 to 100.0]
  Day 14 (n=101) | 99.0 [94.3 to 100.0]
  Day 28 (n=102) | 95.9 [89.9 to 98.9]

4. Secondary Outcome: Mycological Efficacy: Eradication Rate
Description: Determined based on the results of culture of Candida as Eradication, Persistent or Indeterminate.
  Eradication rate was calculated based on the following formula, "the number of participants assessed as Eradication" over "total participants excluding ones assessed as Indeterminate" multiplied by 100.
Time Frame: Day 7, Day 14 and Day 28
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fluconazole
Number analyzed (Participants) | 102
percentage of participants
  Day 7 (n=95) | 95.7 [89.5 to 98.8]
  Day 14 (n=100) | 89.8 [82.0 to 95.0]
  Day 28 (n=102) | 85.9 [77.4 to 92.0]

5. Secondary Outcome: Total Scores for Clinical Symptoms
Description: Sum of severity scores in vulvovaginal itching, vulvovaginal burning sensation, excoriation of vulva, vaginal discharge, vulva oedema, redness of vulva, vaginal redness, property of vaginal content. Higher scores show greater severity. Total Scores for Clinical Symptoms Severity range from 0 (best possible outcome) to 24 (worst possible outcome).
Time Frame: Day 1 (before dosing), Day 3, Day 7, Day 14 and Day 28
Population: as for outcome 1
Measure: Mean (Full Range); unit: score on s scale
Arm/Group | Fluconazole
Number analyzed (Participants) | 102
score on s scale
  Day 1 (before dosing, n=102) | 11.0 [4 to 19]
  Day 3 (n=98) | 4.5 [0 to 12]
  Day 7 (n=93) | 1.8 [0 to 10]
  Day 14 (n=98) | 0.8 [0 to 7]
  Day 28 (n=99) | 0.4 [0 to 9]

6. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: Before dosing and 2, 24, 48 and 168 hours after dosing
Population: The plasma parameter analysis set was defined as those participants who were included in the plasma concentration analysis set and for whom at least one set of plasma concentration parameters was calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Fluconazole
Number analyzed (Participants) | 157
mcg/mL | 3.71 (24)

7. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: Before dosing and 2, 24, 48 and 168 hours after dosing
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | Fluconazole
Number analyzed (Participants) | 157
hours | 1.9 [1.8 to 70.3]

8. Secondary Outcome: Area Under the Plasma Curve From Time Zero to Last Quantifiable Concentration (AUClast)
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Time Frame: Before dosing and 2, 24, 48 and 168 hours after dosing
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*h/mL
Arm/Group | Fluconazole
Number analyzed (Participants) | 149
mcg*h/mL | 156.1 (22)

9. Secondary Outcome: Maximum Observed Concentration (Cmax) for Vaginal Fluid Fluconazole Concentration Adjusted by Sample Weight
Time Frame: Before dosing and 2, 24, 48 and 168 hours after dosing
Population: The vaginal discharge parameter analysis set was defined as those participants who were included in the vaginal discharge concentration analysis set and for whom at least one set of vaginal discharge parameters was calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/g
Arm/Group | Fluconazole
Number analyzed (Participants) | 157
mcg/g | 1.33 (49)

10. Secondary Outcome: Time to Reach Maximum Observed Concentration (Tmax) for Vaginal Fluid Fluconazole Concentration Adjusted by Sample Weight
Time Frame: Before dosing and 2, 24, 48 and 168 hours after dosing
Population: as for outcome 9
Measure: Median (Full Range); unit: hours
Arm/Group | Fluconazole
Number analyzed (Participants) | 157
hours | 20.5 [1.8 to 116.6]

11. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for Vaginal Fluid Fluconazole Concentration Adjusted by Sample Weight
Description: Area under the concentration time-curve from zero to the last measured concentration (AUClast) for Vaginal Fluid Fluconazole Concentration adjusted by Sample Weight
Time Frame: Before dosing and 2, 24, 48 and 168 hours after dosing
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*h/g
Arm/Group | Fluconazole
Number analyzed (Participants) | 144
mcg*h/g | 79.5 (43)

12. Secondary Outcome: Maximum Observed Concentration (Cmax) for Vaginal Fluid Fluconazole Concentration Adjusted by Potassium in Vaginal Fluid
Time Frame: Before dosing and 2, 24, 48 and 168 hours after dosing
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Fluconazole
Number analyzed (Participants) | 157
mcg/mL | 1.53 (59)

13. Secondary Outcome: Time to Reach Maximum Observed Concentration (Tmax) for Vaginal Fluid Fluconazole Concentration Adjusted by Potassium in Vaginal Fluid
Time Frame: Before dosing and 2, 24, 48 and 168 hours after dosing
Population: as for outcome 9
Measure: Median (Full Range); unit: hrs
Arm/Group | Fluconazole
Number analyzed (Participants) | 157
hrs | 20.5 [1.8 to 116.6]

14. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for Vaginal Fluid Fluconazole Concentration Adjusted by Potassium in Vaginal Fluid
Description: Area under the concentration time-curve from zero to the last measured concentration (AUClast) for Vaginal Fluid Fluconazole Concentration Adjusted by Potassium in Vaginal Fluid
Time Frame: Before dosing and 2, 24, 48 and 168 hours after dosing
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*h/mL
Arm/Group | Fluconazole
Number analyzed (Participants) | 142
mcg*h/mL | 85.3 (48)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Fluconazole
Serious Adverse Events (participants affected / at risk) | 0/157
Other Adverse Events (participants affected / at risk) | 37/157
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluconazole (N=157)
Palpitations (Cardiac disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Pyrexia (General disorders) | 2
Bronchitis (Infections and infestations) | 2
Bronchopneumonia (Infections and infestations) | 1
Chlamydial infection (Infections and infestations) | 1
Cystitis (Infections and infestations) | 4
Folliculitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Genital herpes (Infections and infestations) | 4
Nasopharyngitis (Infections and infestations) | 8
Pharyngitis streptococcal (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Vulvovaginitis trichomonal (Infections and infestations) | 1
Burns first degree (Injury, poisoning and procedural complications) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Genital haemorrhage (Reproductive system and breast disorders) | 3
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 4
Urticaria (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.